CLINICAL TRIAL: NCT00243581
Title: The Effects of an Intensive Lifestyle Modification Program on Carotid Artery Intima-Media Thickness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SwedishAmerican Health System (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: SACCM Ornish Clinical Trial
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Last update posted 2005-10-31 (Estimated); Status verified 2005-05

CONDITIONS: a Myocardial Infarction; Coronary Artery Bypass Graft Surgery Percutaneous Transluminal Coronary Angioplasty Stent Placement

INTERVENTIONS:
Behavioral: Dean Ornish Heart Disease Reversing Program

SUMMARY:
The objective of this study is to evaluate the effect of the Ornish Program on cardiovascular disease as measured by the IMT of the common carotid artery, and to compare this effect to outcomes from patients participating in traditional cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

Patients will be accepted into the study if they demonstrate one or more of the following within the previous 12 months: a myocardial infarction, coronary artery bypass graft surgery, or percutaneous transluminal coronary angioplasty, stent placement, or rotoblator procedures. Patients will also accepted if they have stable angina as determined by the Rose Questionnaire or pacemaker associated with one or more of the previously mentioned diagnoses. For the purposes of this study, myocardial infarction is defined as the presence of at least two of the following three criteria: continuous chest pain lasting at least 30 minutes; electrocardiogram changes expressing an evolving myocardial infarction (ST segment elevation or depression, evolving Q waves, or symmetric inversion of T waves); or elevated cardiac enzyme levels (at least twice the I levels).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Steven G. Aldana, Ph.D., Principal Investigator — SwedishAmerican Health System